CLINICAL TRIAL: NCT05797909
Title: The PCOS Challenge Study: For the Collection of Information to Advance Research and Improve Care for PCOS Patients
Brief Title: The PCOS Challenge Study
Acronym: PCOSCHALLENGE
Status: Recruiting | Type: Observational
Sponsor: PCOS Challenge: The National Polycystic Ovary Syndrome Association (Other)
Responsible Party: Sponsor
Other Study IDs: PCOSC001
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: pcos; polycystic ovary syndrome; polycystic ovarian syndrome; stein leventhal syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Target Population: The target population includes individuals diagnosed with PCOS by a healthcare provider, self-diagnosed with PCOS, or who are exhibiting PCOS Symptoms and willing to sign the consent.
- Control Population: The control population includes people born biologically female who have not been diagnosed with PCOS and who also do not have symptoms of PCOS.

SUMMARY:
The primary purpose of The PCOS Challenge Study will be to conduct high-quality research where patients are included in the design, and answering the questions that patients identify as important to their lived experience with PCOS. In partnership with clinical investigators, patients will work on the development and management of data collection, the research agenda, and the sharing of research findings. The PCOSC Study will promote the advancement of research that provides reliable, useful, and meaningful information to patients with PCOS and their clinicians.

The population for The PCOS Challenge Study will include individuals with a clinical diagnosis of PCOS, individuals self-diagnosed with PCOS, individuals with symptoms of PCOS (e.g., hirsutism, irregular menstrual cycles), and demographic-matched controls without PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PCOS by a health professional, self-diagnosed with PCOS or individuals with PCOS symptoms
* Willing to sign the consent form
* Able to understand the registry surveys or what is being asked

Exclusion Criteria:

* Unable to understand the surveys or what is being asked
* Unwilling to sign the consent form

Ages: 12 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Born biologically female
Study Population: The population for The PCOS Challenge Study will include individuals with a clinical diagnosis of PCOS, individuals self-diagnosed with PCOS, individuals with symptoms of PCOS (e.g., hirsutism, irregular menstrual cycles), and demographic-matched controls without PCOS.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2042-06 (Estimated); Study Completion 2042-12-31 (Estimated)

PRIMARY OUTCOMES:
Information | One Year
  Such as responses to survey questions

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Ottey, MHA, MT (ASCP), Principal Investigator — PCOS Challenge: The National Polycystic Ovary Syndrome Association; Ricardo Azziz, MD, MPH, MBA, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- PCOS Challenge: The National Polycystic Ovary Syndrome Association, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in PCOS. Data or samples shared will be coded, with no PHI included.
Supporting Information: Study Protocol